CLINICAL TRIAL: NCT01259050
Title: Phase 1 Open Label Study of Zinc Therapy in ALS Patients
Brief Title: Safety Study of High Doses of Zinc in ALS Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Phoenix Neurological Associates, LTD (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Zinc-ALS
Record Dates: First submitted 2010-12-10; First posted 2010-12-13 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-03

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS treatment; Zinc; Copper; BMAA; ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Zinc; Copper

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Zinc and Copper (Experimental)
  Interventions: Drug: Zinc and Copper

INTERVENTIONS:
Drug: Zinc and Copper — Optizinc 90 mg/d Copper 1 mg

SUMMARY:
The purpose of this study is to determine the safety of Zinc given at 90mg/d in conjunction with 2mg/d of copper in ALS patients.

DETAILED DESCRIPTION:
Physicians at Phoenix Neurological Associates (PNA) are looking for individuals diagnosed with ALS to participate in an open label phase II safety trial with zinc in conjunction with copper, used in combination with Riluzole for treating ALS. This investigator initiated trial conducted by Drs. Todd Levine and David Saperstein will help determine if zinc given at high doses is safe and tolerated and could possibly slow the progression of ALS.

Over fifty years ago an epidemic of ALS was discovered on the Island of Guam where a disease complex of ALS was found to be one hundred times more prevalent than in the rest of the world. Research on ALS in Guam linked ALS, along with Parkinson's Disease and Dementia, with a neurotoxin, β-methylamino-L-alanine (BMAA). BMAA is a non-essential amino acid and is produced by a cyanobacterium found in large concentrations in the food consumed by the people on Guam. Subsequently several groups have identified high concentrations of BMAA in brain tissues of patients from North America and Europe with several neurodegenerative diseases including ALS, Parkinson's Disease and Alzheimer's Diseases.

A small proportion of ALS, (about 2%), is associated with a mutation in the superoxide dismutase (SOD1) gene. Mice who express this mutant gene exhibit a progressive, ALS-like neurodegenerative disease.Since it is known that SOD1 binds zinc, and many of the mutant forms of this enzyme associated with ALS show altered zinc binding, zinc may play a key role in all pathological processes associated with ALS. Previous studies have shown that in ALS mutant G93A SOD transgenic mice, actual zinc supplementation delayed death. Zinc has also been thought to serve as an endogenous antioxidant in the central nervous system and help protect the BBB against oxidative stress and prevent BMAA from crossing into the brain.

It has been demonstrated that BMAA binds exceptionally strongly to transition metal ions such as zinc, copper, and nitrogen. If BMAA crossed over the permeable BBB, and enters a compartment in which glutamate was bound to zinc, then the glutamate/zinc complex would dissociate in favor of zinc having a stronger affinity to BMAA. This could lead to higher levels of unbound glutamate which is believed to be highly neurotoxic in ALS patients. We hypothesize by exposing patients to high levels of zinc, both BMAA and glutamate would be kept in a bound complex with zinc, i.e. eliminating competitive binding for zinc, which lead to less excitotoxic free glutamate and glutamate toxicity would be reduced.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-85
2. Male or Female
3. Clinically definite or probable ALS by El Escorial criteria
4. ALS-FRS > 25
5. If on Riluzole they must be on a stable dose for at least 30 days prior to screening
6. Capable of providing informed consent and complying with trial procedures

Exclusion Criteria:

1. Patients with FVC below 50%
2. History of liver disease
3. Severe renal failure
4. Creatinine greater than or equal to 1.5 mg/dL
5. History of intolerance to zinc or copper
6. Evidence of motor neuron disease for greater than 5 years
7. Any other co-morbid condition which would make completion of the trial unlikely
8. If female, pregnant or breast-feeding; or, if of childbearing age, an unwillingness to use birth control.
9. Any other trial medications. Non-trial medications are not cause for exclusion
10. Patient with history of significant anemia
11. Elevated levels of zinc at baseline
12. Patients with copper levels below normal at baseline

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of high doses of zinc in patients with ALS | 1 year

SECONDARY OUTCOMES:
Measure levels of BMAA in blood and urine to determine if there is a decline in these levels over the course of treatment | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Todd D Levine, MD, Principal Investigator — Phoenix Neurological Associates, LTD; David S Saperstein, MD, Principal Investigator — Phoenix Neurological Associates, LTD
Locations (1):
- Phoenix Neurological Associates, Phoenix, Arizona, United States